CLINICAL TRIAL: NCT03645707
Title: A Mixed Methods Evaluation of a Resilience Intervention With Psychoeducational Sessions for Critical Care Nurses
Brief Title: Resilience Insight Self Compassion and Empowerment (RISE) Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1256670
Record Dates: First submitted 2018-08-21; First posted 2018-08-24 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Stress
Keywords: Critical Care Nurse; Resilience; Stress Mindset

STUDY DESIGN:
Intervention Model Description: This is a secondary study to the primary study titled "A Randomized Controlled Trial of a Resilience Intervention for Critical Care Nurses" (Florida Hospital IRBNet #1234568). In the primary study, participants will be randomized into the intervention group or wait-list control group. However, in this secondary study, all participants will attend the 1-day CAR Training Program and the follow-up psychoeducational group sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR Training and Psychoeducational Sessions (Experimental): This is a secondary study to the primary study titled "A Randomized Controlled Trial of a Resilience Intervention for Critical Care Nurses" (IRBNet #1234568). In the primary study, participants will be randomized into the intervention group or wait-list control group.
  In this secondary study, all participants will attend the 1-day CAR Training Program and the follow-up psychoeducational group sessions.
  Interventions: Behavioral: CAR Training and Psychoeducational Sessions

INTERVENTIONS:
Behavioral: CAR Training and Psychoeducational Sessions — Participation in the CAR Training Program, a 1-day training program developed by the J&J Human Performance Institute (HPI). The CAR Training Program uses a holistic approach that focuses on moving between stress and strategic recovery to help build resilience and enable higher performance.
  Participants will attend eight weekly follow-up psychoeducational group sessions facilitated by a licensed mental health counselor that will meet for 90 minutes. The themes of these sessions will be RISE - Resilience, Insight, Self-Compassion, and Empowerment. Due to limited time and flexibility in sessions, participants will practice skills through optional homework activities to facilitate learning between sessions.

SUMMARY:
The purpose of this pilot study is to determine whether the combination of the Corporate Athlete® Resilience (CAR) Training Program and follow-up psychoeducational group sessions has significant impact on nurses' resilience and stress mindset in their personal lives and their working environment. Knowledge from this study can be applied to interventions in the future to improve resilience behavior.

DETAILED DESCRIPTION:
The ongoing nursing shortage in the U.S health care system is a multifaceted issue. One factor leading to the nursing shortage is high turnover, particularly among critical care nurses due to their experiences with stressful work environments, ethical dilemmas, and high rates of patient morbidity and mortality. There is also a high prevalence of psychological disorders, such as anxiety, depression, and Post Traumatic Stress Disorder (PTSD) among critical care nurses. Consequences of turnover and low nurse staffing include lower quality of care, lower patient satisfaction, increased medical errors, increased rates of health care associated infections, and higher 30-day mortality rates.

Resilience is defined as "the ability to adapt to life's ever-changing landscape and recover quickly from the stressors and potential stressors". It is a learned psychological characteristic that can be used to bounce back after disruption and successfully adapt to stressful work experiences in a positive manner.

The Corporate Athlete® Resilience (CAR) Training Program is a 1-day training program that uses a holistic approach that focuses on moving between stress and strategic recovery to help build resilience and enable higher performance.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥ 18 years old.
2. Employed as a critical care nurse at Florida Hospital in an adult ICU, PICU, PCVICU, or Level 3 NICU.
3. Able to speak, read, and understand English fluently.
4. Able to provide informed consent.
5. Receive a high score of ≥ 27 on the Emotional Exhaustion domain and/or a high score of ≥ 13 on the Depersonalization domain of the Maslach Burnout Inventory (MBI) as part of Florida Hospital IRBNet #1234568.
6. Willing to attend a full-day training program at HPI on the designated training date.
7. Willing and able to comply with all study procedures and requirements for the duration of the study.

Exclusion Criteria:

1. At imminent risk of harm to themselves or others

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Stress Mindset Measure - General (SMM-G) | Change from Baseline SMM-G score at 6-months post CAR Training
  Participants will respond to an 8-item questionnaire measuring stress. Responses will be provided on the following 5-point scale: 0=Strongly Disagree, 1=Disagree, 2=Neither Agree nor Disagree, 3=Agree, 4=Strongly Agree.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | Change from Baseline PSS score at 6-months post CAR Training
  Participants will respond to a 10-item questionnaire measuring perceived stress. Responses will be provided on the following 5-point scale: 0=Never, 1=Almost Never, 2=Sometimes, 3=Fairly Often, 4=Very Often.
Brief Resilience Scale (BRS) | Change from Baseline BRS score at 6-months post CAR Training
  Participants will respond to a 6-item questionnaire measuring resilience. Responses will be provided on the following 5-point scale: 1=Strongly Disagree, 2=Disagree, 3=Neutral, 4=Agree, 5=Strongly Agree.
Maslach Burnout Inventory Human Services Survey (MBI-HSS) for Medical Personnel (MP) | Change from Baseline MBI-HSS (MP) score at 6-months post CAR Training
  Participants will respond to a 22-item questionnaire measuring burnout. Responses will be provided on the following 7-point scale: 0=Never, 1=A few times a year or less, 2=Once a month or less, 3=A few times a month, 4=Once a week, 5=A few times a week, 6=Everyday.
Public Health Surveillance - Wellbeing Scale (PHS-WB) | Change from Baseline PHS-WBscore at 6-months post CAR Training
  Participants will respond to a 10-item questionnaire measuring perception of personal well-being and satisfaction. Responses will be provided on a 5-point scale (6 items) and a 10-point scale (4 items).
RAND Medical Outcomes Study (MOS) Sleep Scale Survey | Change from Baseline RAND MOS Sleep Scale score at 6-months post CAR Training
  Participants will respond to a 12-item questionnaire with self-reported information related to sleep patterns. Responses will be provided on the following 6-point scale: 1=All of the time, 2=Most of the time, 3=A good bit of the time, 4=Some of the time, 5=A little of the time, 6=None of the time.
RAND 36-Item Short Form Health Survey (SF-36) | Change from Baseline SF-36 score at 6-months post CAR Training
  Participants will respond to a 36-item questionnaire with self-reported health ratings and perceived impact of one's health on a variety of daily activities. Response options for questionnaire items vary from 3-point scale, 5-point scale, and Yes/No responses.
Absenteeism and Presenteeism questions of the World Health Organization's Health and Work Performance Questionnaire (WHO-HPQ) | Change from Baseline WHO-HPQ score at 6-months post CAR Training
  Participants will respond to 11 absenteeism and presenteeism questions abstracted from the full HPQ. Responses for 2 items require self-reported information regarding hours worked and hours the employer expects the participant to work in 7 days. 6 items require participants to provide work experience information from the past 4 weeks. Responses for 3 items are provided on a 10-point scale in which 0=Worst Performance, and 10=Top Performance. Responses are input into a provided formula for scoring; a higher absenteeism score indicates higher amount of absenteeism, while a higher presenteeism score indicates lower amount of lost performance.
Work Productivity and Activity Impairment Questionnaire (WPAI) | Change from Baseline WPAI score at 6-months post CAR Training
  Participants will respond to a 6-item questionnaire, answering questions about the perceived effect of personal health problems on one's ability to work or perform activities. Responses are provided in a Yes/No format or using a 10-point scale in which 0=Health problems had no effect on my work and 10=Health problems completely prevented me from working.
Self-Reflection and Insight Scale (SRIS) | Change from Baseline SRIS score at 6-months post CAR Training
  Participants will respond to a 20-item questionnaire using a 6-point scale where 1=Strongly disagree and 6=Strongly agree.
Self-Compassion Scale - Short Form (SCS-SF) | Change from Baseline SCS-SF score at 6-months post CAR Training
  Participants will respond to a 12-item questionnaire, indicating how often certain behaviors are personally experienced when in difficult times. Responses are provided on 5-point scale in which 1=Almost never and 5=Almost always.
Psychological Empowerment Instrument | Change from Baseline Psychological Empowerment Instrument score at 6-months post CAR Training
  Participants will respond to a 12-item questionnaire to items regarding self-orientations people may have with regard to their work role. Responses are provided on the following 7-point scale: 1=Very strongly disagree, 2=Strongly disagree, 3=Disagree, 4=Neutral, 5=Agree, 6=Strongly Agree, 7=Very Strongly Agree.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda T. Sawyer, PhD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Acker KH. Do critical care nurses face burnout, PTSD, or is it something else?: getting help for the helpers. AACN Clin Issues Crit Care Nurs. 1993 Aug;4(3):558-65. PMID 8136229
- [Background] Bann CM, Kobau R, Lewis MA, Zack MM, Luncheon C, Thompson WW. Development and psychometric evaluation of the public health surveillance well-being scale. Qual Life Res. 2012 Aug;21(6):1031-43. doi: 10.1007/s11136-011-0002-9. Epub 2011 Sep 23. PMID 21947657
- [Background] Hughes RG, editor. Patient Safety and Quality: An Evidence-Based Handbook for Nurses. Rockville (MD): Agency for Healthcare Research and Quality (US); 2008 Apr. Available from http://www.ncbi.nlm.nih.gov/books/NBK2651/ PMID 21328752
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Crum AJ, Salovey P, Achor S. Rethinking stress: the role of mindsets in determining the stress response. J Pers Soc Psychol. 2013 Apr;104(4):716-33. doi: 10.1037/a0031201. Epub 2013 Feb 25. PMID 23437923
- [Background] Grant, A. M., Franklin, J., & Langford, P. (2002). The Self-Reflection and Insight Scale: A new measure of private self-consciousness. Social Behavior and Personality, 30(8), 821-836.
- [Background] Johnson & Johnson Health & Wellness Solutions Research Team. 2017. Validation and Analysis of Johnson & Johnson Human Performance Institute™ (HPI) Assessment Inventory. Unpublished manuscript.
- [Background] Kessler RC, Barber C, Beck A, Berglund P, Cleary PD, McKenas D, Pronk N, Simon G, Stang P, Ustun TB, Wang P. The World Health Organization Health and Work Performance Questionnaire (HPQ). J Occup Environ Med. 2003 Feb;45(2):156-74. doi: 10.1097/01.jom.0000052967.43131.51. PMID 12625231
- [Background] Maslach, C., Jackson, S. E., & Leiter, M. P. (1996). Maslach Burnout Inventory manual (3rd ed.). Palo Alto, CA: Consulting Psychologists Press.
- [Background] Mealer ML, Shelton A, Berg B, Rothbaum B, Moss M. Increased prevalence of post-traumatic stress disorder symptoms in critical care nurses. Am J Respir Crit Care Med. 2007 Apr 1;175(7):693-7. doi: 10.1164/rccm.200606-735OC. Epub 2006 Dec 21. PMID 17185650
- [Background] Mealer M, Burnham EL, Goode CJ, Rothbaum B, Moss M. The prevalence and impact of post traumatic stress disorder and burnout syndrome in nurses. Depress Anxiety. 2009;26(12):1118-26. doi: 10.1002/da.20631. PMID 19918928
- [Background] Mealer M, Conrad D, Evans J, Jooste K, Solyntjes J, Rothbaum B, Moss M. Feasibility and acceptability of a resilience training program for intensive care unit nurses. Am J Crit Care. 2014 Nov;23(6):e97-105. doi: 10.4037/ajcc2014747. PMID 25362680
- [Background] Mealer M, Jones J, Newman J, McFann KK, Rothbaum B, Moss M. The presence of resilience is associated with a healthier psychological profile in intensive care unit (ICU) nurses: results of a national survey. Int J Nurs Stud. 2012 Mar;49(3):292-9. doi: 10.1016/j.ijnurstu.2011.09.015. Epub 2011 Oct 5. PMID 21974793
- [Background] Pipe TB, Buchda VL, Launder S, Hudak B, Hulvey L, Karns KE, Pendergast D. Building personal and professional resources of resilience and agility in the healthcare workplace. Stress Health. 2012 Feb;28(1):11-22. doi: 10.1002/smi.1396. Epub 2011 Mar 13. PMID 22259154
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] RAND Corporation. (2018). Sleep Scale Survey. Retrieved from https://www.rand.org/health/surveys_tools/mos/sleep-scale.html.
- [Background] RAND Corporation. (2018). 36-Item Short Form Survey (SF-36). Retrieved from https://www.rand.org/health/surveys_tools/mos/36-item-short-form.html.
- [Background] Reilly MC, Zbrozek AS, Dukes EM. The validity and reproducibility of a work productivity and activity impairment instrument. Pharmacoeconomics. 1993 Nov;4(5):353-65. doi: 10.2165/00019053-199304050-00006. PMID 10146874
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Spreitzer, G. M. (1995). Psychological empowerment in the workplace: Dimensions, measurement, and validation. Academy of Management Journal, 38(5), 1442-1465.